CLINICAL TRIAL: NCT03603964
Title: An Open-Label, Multicenter, Extension Study for Subjects Who Participated in Prior Guadecitabine Clinical Studies
Brief Title: Guadecitabine Extension Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination not due to patient safety
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGI-110-12
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Results first posted 2023-04-26 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia; Myeloid Dysplastic Syndrome
Keywords: Guadecitabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Guadecitabine (Experimental): Participants received guadecitabine, subcutaneous (SC) injection on Days 1-5 of each 28-day cycle at the same dose that they were receiving in the last cycle of their prior study or at a different dose as guided by the dose adjustment guidelines in the prior study protocol.
  Interventions: Drug: Guadecitabine

INTERVENTIONS:
Drug: Guadecitabine — Guadecitabine
  Other Names: SGI-110

SUMMARY:
This is a multicenter, open-label extension study for participants who participated in a previous Astex-sponsored guadecitabine clinical study [including but not limited to SGI-110-01 (NCT01261312), SGI-110-04 (NCT02348489), SGI-110-06 (NCT02920008), and SGI-110-07 (NCT02907359)].

DETAILED DESCRIPTION:
Participants who were still receiving treatment with guadecitabine and in the opinion of the investigator were still benefitting from treatment at the time of database close of the original study will be eligible to participate in this extension study. Approximately 250 subjects could be enrolled.

Participants will attend clinic visits on Days 1-5 of each 28-day cycle to receive treatment with guadecitabine. Data collection will be limited to treatment exposure, adverse events, concomitant medications, limited laboratory parameters, and survival status.

ELIGIBILITY:
Inclusion Criteria:

1. Previous participation in an Astex-sponsored guadecitabine clinical trial [including but not limited to SGI-110-01 (NCT01261312), SGI-110-04 (NCT03603964), SGI-110-05, SGI-110-06 (NCT02920008), and SGI-110-07 (NCT02907359)], in which the participant was treated with guadecitabine and was still on active treatment with guadecitabine at the time of database close for the prior study.
2. Participant is considered to be benefitting from guadecitabine treatment in the opinion of the treating investigator.
3. Able to understand and comply with the study procedures, understand the risks involved in the study, and provide written informed consent before any study-specific procedure.
4. Women of child-bearing potential (according to recommendations of the Clinical Trial Facilitation Group [CTFG]) must not be pregnant or breastfeeding and must have a negative pregnancy test at screening. Women of child-bearing potential and men with female partners of child-bearing potential must agree to practice 2 highly effective contraceptive measures while receiving treatment with guadecitabine and for at least 3 months after completing treatment and must agree not to become pregnant or father a child while receiving study treatment and for at least 3 months after completing guadecitabine treatment.

Exclusion Criteria:

* 1. Any participant who, in the opinion of the investigator, may have other conditions, organ dysfunction, or have safety data from their prior study participation that suggest that the risks of continuing treatment with guadecitabine may outweigh the benefits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (5):
  - Roswell Park, Buffalo, New York
  - Duke Cancer Center, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - Center for Blood Cancers, Nashville, Tennessee
- Medizinische Universität Graz, Graz, Styria, Austria
- Canada (2):
  - The Ottawa Hospital - General, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
- Rigshospitalet-Copenhagen University Hospital, Copenhagen, Denmark
- Italy (4):
  - Azienda Ospedaliera SS. Antonio E. Biagio E. Cesare Arrigo di Alessandria, Alessandria
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliero Universitaria S. Maria della Misericordia di Udine, Udine
- Japan (3):
  - Tokai University Hospital, Isehara-shi
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - Saga University Hospital, Saga
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Ulsan University Hospital, Ulsan
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Taiwan (2):
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 32 study centers in the United States, Spain, Italy, Canada, Japan, France, Germany, Poland, Finland, South Korea, Taiwan, Czech Republic and Australia from 18 July 2018 to 30 November 2020.
Pre-assignment Details: 35 participants who had participated in a previous Astex-sponsored guadecitabine clinical study (SGI-110-01 {NCT01261312}, SGI-110-04 {NCT02348489}, SGI-110-06 {NCT02920008}, and SGI-110-07 {NCT02907359}) and were still benefitting from the treatment at the time of database close of the original study, were enrolled in this extension study.
Groups:
- Guadecitabine: Participants received guadecitabine, subcutaneous (SC) injection on Days 1-5 of each 28-day cycle at the same dose that they were receiving in the last cycle of their prior study or at a different dose as guided by the dose adjustment guidelines in the prior study protocol up to a maximum of 26 cycles.
Period: Overall Study
Arm/Group | Guadecitabine
Started | 35
Completed | 0
Not Completed | 35
Not completed — Death | 9
Not completed — Withdrawal by participant | 7
Not completed — Study terminated by Sponsor | 19

BASELINE CHARACTERISTICS:
Population: Efficacy population included all participants who received any amount of study treatment.
Groups:
- Guadecitabine: Participants received guadecitabine, SC injection on Days 1-5 of each 28-day cycle, up to at the same dose that they were receiving in the last cycle of their prior study or at a different dose as guided by the dose adjustment guidelines in the prior study protocol up to a maximum of 26 cycles.
Arm/Group | Guadecitabine
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE can therefore be any unfavorable and unintended sign (including a clinically significant abnormal finding in laboratory tests or other diagnostic procedures), symptom, or disease temporally associated with the use of a drug, without any judgment about causality. TEAEs are defined as events that occur or worsen on or after the date of the first study treatment (Cycle 1 Day 1 {C1D1}) until 30 days after the last dose of study treatment or the start of an alternative anti-cancer treatment, whichever occurs first.
Time Frame: From the start of study treatment until 30 days after the last dose of study treatment or prior to the participant receiving alternative anticancer therapy, whichever occurs first.
Population: Safety population included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Guadecitabine
Number analyzed (Participants) | 35
Participants | 31

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the number of days from the time of randomization in the prior study to the date of death (regardless of cause). Participants without a documented death date at the time of analysis were censored at the last date known alive. Survival time in days = (earliest of date of death or censoring) - (randomization date in the prior study).
Time Frame: From randomization in the prior study to the date of death
Population: Efficacy population included all participants who received any amount of study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Guadecitabine
Number analyzed (Participants) | 35
days | 2583.0 [1422.0 to NA] — Not estimable with current data due to early termination.

ADVERSE EVENTS:
Time Frame: From the start of study treatment until 30 days after the last dose of study treatment or prior to the participant receiving alternative anticancer therapy, whichever occurs first.
Description: Safety population included all participants who received any amount of study drug.
Arm/Group | Guadecitabine
All-Cause Mortality (participants affected / at risk) | 9/35
Serious Adverse Events (participants affected / at risk) | 20/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guadecitabine (N=35)
Febrile neutropenia (Blood and lymphatic system disorders) | 7
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 6
Sepsis (Infections and infestations) | 3
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early not due to participant safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/64/NCT03603964/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT03603964/SAP_001.pdf